CLINICAL TRIAL: NCT04557956
Title: Phase 1/2 Study of an EZH2 Inhibitor (Tazemetostat) in Combination With Dual BRAF/MEK Inhibition in Patients With BRAF- Mutated Metastatic Melanoma Who Progressed on Prior BRAF/MEK Inhibitor Therapy
Brief Title: Testing the Addition of the Anti-cancer Drug, Tazemetostat, to the Usual Treatment (Dabrafenib and Trametinib) for Metastatic Melanoma That Has Progressed on the Usual Treatment
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-07044; NCI-2020-07044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 202103077; 10285 (Other: Yale University Cancer Center LAO); 10285 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2020-09-18; First posted 2020-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Biopsy; dabrafenib; Magnetic Resonance Spectroscopy; tazemetostat; trametinib

STUDY DESIGN:
Intervention Model Description: Phase I single-arm trial followed by randomized two-arm phase II trial with cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib) (Experimental): Patients receive tazemetostat PO BID, dabrafenib PO BID, and trametinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy, CT scan, MRI, and MUGA or ECHO throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Computed Tomography; Drug: Dabrafenib Mesylate; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Tazemetostat Hydrobromide; Drug: Trametinib Dimethyl Sulfoxide
- Phase II, Arm 1 (tazemetostat) (Active Comparator): Patients receive tazemetostat PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and MRI throughout the study. At the time of progression, patients may crossover to Arm 2 after completion of radiation therapy.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Tazemetostat Hydrobromide

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
  Arms: Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib)
Drug: Tazemetostat Hydrobromide — Given PO
  Other Names: EPZ-6438 Monohydrobromide; Tazemetostat Monohydrobromide; TAZVERIK
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras
  Arms: Phase I; Phase II Arm 2 (tazemetostat, dabrafenib, trametinib)

SUMMARY:
This phase I/II trial investigates the best dose, possible benefits and/or side effects of tazemetostat in combination with dabrafenib and trametinib in treating patients with melanoma that has a specific mutation in the BRAF gene (BRAFV600) and that has spread from where it first started (primary site) to other places in the body (metastatic). Tazemetostat, dabrafenib, and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving tazemetostat in combination with dabrafenib and trametinib may stabilize BRAFV600 mutated melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify a maximum tolerated dose for the EZH2 inhibitor, tazemetostat hydrobromide (tazemetostat), when used in combination with dual BRAF inhibitor (dabrafenib mesylate [dabrafenib]) and MEK inhibitor (trametinib dimethyl sulfoxide [trametinib]) therapy in BRAF/MEK inhibitor-resistant, BRAF^V600-mutated metastatic melanoma. (Phase 1) II. To determine if the addition of the EZH2 inhibitor, tazemetostat, to BRAF and MEK inhibitor therapy improves progression-free survival over single-agent EZH2 inhibitor therapy in patients with BRAF/MEK inhibitor-resistant, BRAF^V600-mutated melanomas harboring an EZH2 alteration. (Phase 2)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase 1) II. To determine the overall response rate of single-agent EZH2 inhibitor therapy (tazemetostat) and triplet EZH2 inhibitor (tazemetostat), BRAF inhibitor (dabrafenib) and MEK inhibitor (trametinib) therapy in patients with BRAF/MEK inhibitor-resistant BRAF^V600-mutated melanomas harboring an EZH2 alteration. (Phase 2)

EXPLORATORY OBJECTIVE:

I. To explore alterations in the gene expression profile (ribonucleic acid [RNA]-sequencing), H3K27 methylome (immunohistochemistry [IHC], chromatin immunoprecipitation [ChIP]-Sequencing), and open chromatin landscape (assay for transposase accessible chromatin [ATAC]-sequencing) with EZH2 inhibition in fresh clinical or patient derived xenograft (PDX)-derived tumor samples, which may reveal underlying transcriptional/epigenetic pathways mediating response to treatment.

OUTLINE: This is a phase I, dose-escalation trial of tazemetostat followed by a phase II trial. Patients in the phase I trial receive treatment as in Arm 2. Patients in the phase II trial are randomized to Arm 1 or Arm 2.

ARM 1: Patients receive tazemetostat orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan and magnetic resonance imaging (MRI) throughout the study. At the time of progression, patients may crossover to Arm 2 after completion of radiation therapy.

ARM 2: Patients receive tazemetostat PO BID, dabrafenib PO BID, and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy, CT scan, MRI, and multigated acquisition scan (MUGA) or echocardiography (ECHO) throughout the study.

After completion of study treatment, patients are followed up at 30 days, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of BRAF^V600E/K-mutated metastatic melanoma
* Patient must have had documented radiographic or clinical evidence of progressive disease while on combination BRAF/MEK inhibitor therapy. For Phase 2 only, no more than one intervening therapy since progression on BRAF/MEK inhibitor therapy is allowed. Subjects who have evidence of progression while on, or within 4 weeks of completing, combination BRAF/MEK inhibitor therapy in the adjuvant setting will be eligible
* PHASE 2 ONLY: Patient must have EZH2 alteration (somatic mutation or copy number alteration). Can be performed on either archival or fresh specimen. EZH2 alterations need to be documented by a Clinical Laboratory Improvement Act (CLIA)/Clinical Laboratory Improvement Program (CLIP)-certified next generation sequencing platform (Foundation One, Tempus, Guardant360, etc.)
* PHASE 2 ONLY: Patient must have measurable disease
* PHASE 2 ONLY: Patient must have at least one tumor lesion amenable to biopsy. If possible, this lesion should be different from the lesion used for following tumor measurements but is not required
* PHASE 2 ONLY: Patient must agree to planned pre-treatment and planned on-treatment biopsy. A pre-treatment biopsy will be optional if patient has an archival tissue block or 5 formalin-fixed paraffin-embedded (FFPE) slides available from specimen used to document presence of eligible EZH2 alteration that is deemed adequate for evaluation
* Patient must be >= 18 years

  * Because no dosing or adverse event data are currently available on the use of tazemetostat in combination with dabrafenib and trametinib in patients < 18 years of age, children are excluded from this study
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Patients with symptomatic central nervous system (CNS) metastases are eligible if previously treated with surgery and/or radiation with no evidence of radiologic CNS recurrence or progression for 4 weeks and on a stable/tapering dose of steroid for at least one week prior to start of study drug. Patients with new or progressive asymptomatic CNS metastases are eligible
* Hemoglobin >= 9 g/dL
* Albumin >= 2.5 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) except subjects with known Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2
* Patients with a prior (or concurrent, if enrolling in Phase 1) malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.3 x institutional ULN. Prophylactic low dose warfarin may be given to maintain central catheter patency
* The effects of tazemetostat, and the combination of tazemetostat, dabrafenib and trametinib on the developing human fetus are unknown. Women of childbearing potential and all male patients must agree to the following:

  * For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period, for 6 months after tazemetostat discontinuation, or for 6 months after discontinuation of the combination of tazemetostat, dabrafenib and trametinib. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately

    * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
    * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
    * Due to the potential of enzyme induction with tazemetostat, female subjects who use hormonal contraceptives should use an additional barrier method of birth control while on study treatment and for 6 months after discontinuation of tazemetostat or the combination of tazemetostat, dabrafenib and trametinib
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception
  * Women of childbearing potential must have a negative urine or serum pregnancy test at screening
  * For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

    * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of study drug. Men must refrain from donating sperm during this same period. In addition, female partners of male subjects should adhere to the following:

      * Intrauterine device (IUD) (must provide medical documentation of IUD)
      * Hormonal contraceptive (partner must be on a stable dose of the same hormonal contraceptive product for at least 4 weeks before receiving study drug) AND a condom (hormonal contraceptives must be supplemented with condoms)
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Have progressed on, been intolerant to, is ineligible for, or has refused prior standard of care anti-PD-1 based immunotherapy

Exclusion Criteria:

* Previous therapy with a demethylating agent (i.e. decitabine) or previous therapy with an EZH2 inhibitor
* History of second malignancy not treated with curative intent
* History of life-threatening toxicity, including hypersensitivity, related to BRAF or MEK inhibitor therapy, or known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Active infection requiring intravenous therapy
* Presence of untreated or progressive symptomatic CNS melanoma metastases. Diffuse leptomeningeal carcinomatosis or metastases causing spinal cord compression are exclusionary. Previously treated lesions should be stable for >= 4 weeks (must be documented by imaging). Subjects on a stable dose of corticosteroids for > 1 week can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for > 4 weeks
* Radiation therapy in the last 14 days. Palliative radiation to a localized area without residual toxicity requires a washout of at least 7 days
* Prior systemic anti-cancer therapy (chemotherapy, targeted therapy, immunotherapy, biologic therapy, or vaccine therapy) within the 2 weeks preceding the first dose of study treatment. For Phase 2 only, prior chemotherapy regimens are not permitted
* Use of other investigational drugs within 21 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study treatment and during the study
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) grade 2 or higher from previous anti-cancer therapy, except alopecia and other toxicities that have resolved to grade 1 or well controlled with medical management (i.e.: hypothyroidism, adrenal insufficiency, type 1 diabetes, etc.), at the time of randomization
* Current use of a prohibited medication. Patients must not be treated with any medications or substances that are strong or moderate inhibitors or inducers of CYP3A or strong inhibitors or inducers of CYP2C8 within 14 days prior to the first treatment through the end of the study. Current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib
* A history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (with the exception of cleared HBV and HCV infection, which will be allowed)
* History of interstitial lung disease or pneumonitis
* Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders. Patients on anticoagulation with low molecular weight heparin or low dose warfarin are allowed
* History of myeloid malignancies, including myelodysplastic syndrome (MDS)
* Has abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and multiple primary neoplasms (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and deoxyribonucleic acid (DNA) sequencing
* History of T-lymphoblastic lymphoma (T-LBL)/T-cell acute lymphoblastic leukemia (T-ALL)
* Patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility
* History or evidence of cardiovascular risks including any of the following:

  * QT interval corrected for heart rate using Fridericia's formula (QT corrected by Fridericia [QTcF]) >= 450 msec
  * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to randomization
  * History or evidence of current class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Intra-cardiac defibrillators
  * Abnormal cardiac valve morphology (>= grade 2) documented by ECHO; (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study
  * History or evidence of current clinically significant uncontrolled cardiac arrhythmias; clarification: Subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
  * Left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN) by ECHO or MUGA
  * Known cardiac metastases
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tazemetostat / dabrafenib / trametinib, breastfeeding should be discontinued prior to treatment
* Patients with uncontrolled diabetes
* Patients with a history of retinal vein occlusion (RVO), retinal pigment epithelial detachment (RPED) or other ophthalmologic toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (Phase I) | Up to 30 days
  Data analysis will be descriptive in nature, and will be determined using the standard 3+3 algorithm. Toxicities by grade, number of cycles administered, and response to treatment will be listed for each dose level.
Median progression-free survival (PFS) (Phase II) | At 6 and 12 months
  Median PFS in each arm will be assessed using Kaplan-Meier product limit methods and the randomized arms will be compared using log-rank test (at 0.15 one-sided significance level) when 36 PFS events are observed.

SECONDARY OUTCOMES:
Overall response rates (complete response, partial response) | Up to 3 years
  Assessed by Response Evaluation Criteria in Solid Tumors 1.1, and 95% confidence intervals will be calculated.
Overall survival | Up to 3 years
  Will be estimated in each arm using Kaplan-Meier product limit methods, and its 95% confidence interval will be calculated.
Incidence of adverse events | Up to 3 years
  Toxicity evaluation will be descriptive, and standard toxicity definitions and criteria will be used as outlined in the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The number and percentage of subjects experiencing each type of adverse event will be tabulated by severity. If appropriate, confidence intervals will be used to characterize the precision of the estimate. A complete listing of adverse events will also be tabulated, and will provide details including severity, relationship to treatment, onset, duration, and outcome. Laboratory data measured on a continuous scale will be characterized by summary statistics (mean and standard deviation).

CONTACTS AND LOCATIONS:
Overall Officials: Tanner M Johanns, Principal Investigator — Yale University Cancer Center LAO
Locations (17):
- United States (17):
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm